CLINICAL TRIAL: NCT00825643
Title: A Multicentre, Open Label, Observational 24-week Study to Evaluate Safety of Initiating Insulin Therapy With Levemir® (Insulin Detemir) Once-daily in Oral Antidiabetic Drug-treated Patients With Type 2 Diabetes
Brief Title: Observational Study to Evaluate the Safety of Levemir® in Type 2 Diabetes
Acronym: SOLVE™
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-3714
Record Dates: First submitted 2009-01-20; First posted 2009-01-21 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Insulin detemir
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Start dose and frequency to be prescribed by the physician as a result of a normal clinical evaluation
  Other Names: NN304, Levemir®

SUMMARY:
This study is conducted in Europe, North America and Asia. The aim of this observational study is to evaluate the safety and effectiveness while using Levemir® once daily in combination with oral antidiabetic drugs in type 2 diabetics during 24 weeks under normal clinical practice.

Data from the NN304-3573 study (NCT00740519) will be pooled with data from this study and reported together in the final study report for this study.

ELIGIBILITY:
Inclusion Criteria:

* After the participating physician's decision has been made to initiate once-daily Levemir® therapy, any patient with Type 2 diabetes who is currently treated with diet, exercise and one or more OADs can be offered to participate

Exclusion Criteria:

* Current treatment with insulin
* Known or suspected allergy to Levemir® or excipients
* Children below the age of 6 years
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant within the next 6 months or are not using adequate contraceptive methods (contraceptive measures as required by local law or practice)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from both general and speciality practice settings who have been deemed appropriate to receive Levemir® as new treatment and as part of routine out-patient care by the prescribing physician
Sampling Method: Non-Probability Sample
Enrollment: 18481 (Actual)
Dates: Start 2008-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse drug reactions (SADRs) including major hypoglycaemia | during 24 weeks of treatment

SECONDARY OUTCOMES:
Incidence of all adverse drug reactions (ADRs) | during 24 weeks of treatment
Incidence of major and minor hypoglycaemic events | in the 4 weeks preceding trial start, and at the 12 and 24 week visits
HbA1c and its change from trial start | at the 12 and 24 week visits
Fasting blood glucose (FBG) (average of the self-monitored blood glucose measurements) and its change from trial start | at the 12 and 24 week visits
FBG variability (measured as standard deviation of FBG) and its change from trial start | at the 12 and 24 weeks visits
Body weight and its change from trial start | at the 12 and 24 week visits

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (9):
- Novo Nordisk Investigational Site, Mississauga, Canada
- Novo Nordisk Investigational Site, Beijing, Beijing Municipality, China
- Novo Nordisk Investigational Site, Mainz, Germany
- Novo Nordisk Investigational Site, Kfar Saba, Israel
- Novo Nordisk Investigational Site, Rome, Italy
- Novo Nordisk Investigational Site, Warsaw, Poland
- Novo Nordisk Investigational Site, Paço de Arcos, Portugal
- Novo Nordisk Investigational Site, Madrid, Spain
- Novo Nordisk Investigational Site, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Khunti K, Damci T, Meneghini L, Pan CY, Yale JF; SOLVE Study Group. Study of Once Daily Levemir (SOLVE): insights into the timing of insulin initiation in people with poorly controlled type 2 diabetes in routine clinical practice. Diabetes Obes Metab. 2012 Jul;14(7):654-61. doi: 10.1111/j.1463-1326.2012.01602.x. Epub 2012 Apr 22. PMID 22443213
- [Result] Khunti K, Caputo S, Damci T, Dzida GJ, Ji Q, Kaiser M, Karnieli E, Liebl A, Ligthelm RJ, Nazeri A, Orozco-Beltran D, Pan C, Ross SA, Svendsen AL, Vora J, Yale JF, Meneghini LF; SOLVE Study Group. The safety and efficacy of adding once-daily insulin detemir to oral hypoglycaemic agents in patients with type 2 diabetes in a clinical practice setting in 10 countries. Diabetes Obes Metab. 2012 Dec;14(12):1129-36. doi: 10.1111/j.1463-1326.2012.01665.x. Epub 2012 Aug 30. PMID 22830956
- [Result] Keating GM. Insulin detemir: a review of its use in the management of diabetes mellitus. Drugs. 2012 Dec 3;72(17):2255-87. doi: 10.2165/11470200-000000000-00000. PMID 23110609
- [Result] Ross S, Dzida G, Ji Q, Kaiser M, Ligthelm R, Meneghini L, Nazeri A, Orozco-Beltran D, Pan C, Svendsen AL; SOLVE Study Group. Safety of once-daily insulin detemir in patients with type 2 diabetes treated with oral hypoglycemic agents in routine clinical practice. J Diabetes. 2014 May;6(3):243-50. doi: 10.1111/1753-0407.12091. Epub 2013 Oct 29. PMID 24103141
- [Result] Vora J, Caputo S, Damci T, Orozco-Beltran D, Pan C, Svendsen AL, Solje KS, Khunti K; SOLVE study group. Effect of once-daily insulin detemir on oral antidiabetic drug (OAD) use in patients with type 2 diabetes. J Clin Pharm Ther. 2014 Apr;39(2):136-43. doi: 10.1111/jcpt.12116. Epub 2013 Dec 13. PMID 24329524
- [Result] Pan C, Han P, Ji L, Ji Q, Lu J, Lin J, Liu J, Su B, Shi J, Wang P. Weight-neutral effect of once-daily insulin detemir in Chinese type 2 diabetes patients: subgroup analysis of the SOLVE study. J Diabetes. 2015 Mar;7(2):222-30. doi: 10.1111/1753-0407.12179. Epub 2014 Sep 4. PMID 24909984
- [Result] Dzida G, Karnieli E, Svendsen AL, Solje KS, Hermanns N; SOLVE Study Group. Depressive symptoms prior to and following insulin initiation in patients with type 2 diabetes mellitus: Prevalence, risk factors and effect on physician resource utilisation. Prim Care Diabetes. 2015 Oct;9(5):346-53. doi: 10.1016/j.pcd.2015.01.002. Epub 2015 Jan 30. PMID 25649990
- [Result] Caputo S, Maran A, Mannino D, Morano S, Lastoria G, Nicoziani P. Safety and effectiveness of insulin detemir in combination with oral antidiabetic agents in an outpatient specialist setting: results of the Italian SOLVE observational study. Minerva Endocrinol. 2015 Dec;40(4):249-58. PMID 26551483
- [Result] Morales C, de Luis D, de Arellano AR, Ferrario MG, Lizan L. Cost-Effectiveness Analysis of Insulin Detemir Compared to Neutral Protamine Hagedorn (NPH) in Patients with Type 1 and Type 2 Diabetes Mellitus in Spain. Diabetes Ther. 2015 Dec;6(4):593-610. doi: 10.1007/s13300-015-0143-x. Epub 2015 Nov 20. PMID 26589521
- [Result] Orozco-Beltran D, Pan C, Svendsen AL, Faerch L, Caputo S; SOLVE Study Group. Basal insulin initiation in primary vs. specialist care: similar glycaemic control in two different patient populations. Int J Clin Pract. 2016 Mar;70(3):236-43. doi: 10.1111/ijcp.12776. Epub 2016 Feb 24. PMID 26916450
- [Result] Khunti K, Damci T, Husemoen LL, Babu V, Liebl A. Exploring the characteristics of suboptimally controlled patients after 24weeks of basal insulin treatment: An individualized approach to intensification. Diabetes Res Clin Pract. 2017 Jan;123:209-217. doi: 10.1016/j.diabres.2016.11.028. Epub 2016 Dec 9. PMID 28061430
- [Derived] Pan C, Ji L, Lu J, Yang W, Zhou Z; Chinese SOLVE Study. [Effectiveness and safety of initiation of once-daily insulin detemir in Chinese patients with type 2 diabetes previously treated with different quantities of oral anti-diabetic drugs: subgroup analysis of the Chinese SOLVE Study]. Zhonghua Nei Ke Za Zhi. 2015 Jul;54(7):612-7. Chinese. PMID 26359024
- [Derived] Damci T, Emral R, Svendsen AL, Balkir T, Vora J; SOLVE study group. Lower risk of hypoglycaemia and greater odds for weight loss with initiation of insulin detemir compared with insulin glargine in Turkish patients with type 2 diabetes mellitus: local results of a multinational observational study. BMC Endocr Disord. 2014 Jul 21;14:61. doi: 10.1186/1472-6823-14-61. PMID 25048824
- [Derived] Yale JF, Damci T, Kaiser M, Karnieli E, Khunti K, Liebl A, Baeres FM, Svendsen AL, Ross SA; SOLVE Study Group. Initiation of once daily insulin detemir is not associated with weight gain in patients with type 2 diabetes mellitus: results from an observational study. Diabetol Metab Syndr. 2013 Oct 2;5(1):56. doi: 10.1186/1758-5996-5-56. PMID 24499517
- [Derived] Liebl A, Andersen H, Svendsen AL, Vora J, Yale JF; SOLVE Study Group. Resource utilisation and quality of life following initiation of insulin detemir in patients with type 2 diabetes mellitus. Int J Clin Pract. 2013 Aug;67(8):740-9. doi: 10.1111/ijcp.12133. PMID 23869677
- [Derived] Karnieli E, Baeres FM, Dzida G, Ji Q, Ligthelm R, Ross S, Svendsen AL, Yale JF; SOLVE Study Group. Observational study of once-daily insulin detemir in people with type 2 diabetes aged 75 years or older: a sub-analysis of data from the Study of Once daily LeVEmir (SOLVE). Drugs Aging. 2013 Mar;30(3):167-75. doi: 10.1007/s40266-013-0054-3. PMID 23371395
- [Derived] Liebl A, Wilhelm B, Kaiser M. [Once daily insulin detemir in patients with type 2 diabetes: results of German centers in a 6-month international observational study (SOLVE)]. MMW Fortschr Med. 2012 Dec 17;154 Suppl 4:102-9. German. PMID 23326928
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com